CLINICAL TRIAL: NCT02209753
Title: Phase II, Randomized, Double-blind, Placebo Controlled, Multi-center, Four Week Trial of BIRB 796 BS 5, 10, 20 and 30 mg Oral Tablets Versus Placebo Administered BID in Patients With Moderate to Severe Plaque-type Psoriasis
Brief Title: BIRB 796 BS Versus Placebo in Patients With Moderate to Severs Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.10
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — doramapimod

ARMS (5):
- BIRB 796 BS, low dose (Experimental)
  Interventions: Drug: BIRB 796 BS, low dose
- BIRB 796 BS, medium dose 1 (Experimental)
  Interventions: Drug: BIRB 796 BS, medium dose 1
- BIRB 796 BS, medium dose 2 (Experimental)
  Interventions: Drug: BIRB 796 BS, medium dose 2
- BIRB 796 BS, high dose (Experimental)
  Interventions: Drug: BIRB 796 BS, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIRB 796 BS, low dose
  Arms: BIRB 796 BS, low dose
Drug: BIRB 796 BS, medium dose 1
  Arms: BIRB 796 BS, medium dose 1
Drug: BIRB 796 BS, medium dose 2
  Arms: BIRB 796 BS, medium dose 2
Drug: BIRB 796 BS, high dose
  Arms: BIRB 796 BS, high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The clinical objective of this study was to determine the effect of BIRB 796 BS on pharmacodynamic markers of psoriasis as a measure of efficacy, to determine the population pharmacokinetics of BIRB 796 BS and to determine the safety of BIRB 796 BS over 4 weeks of treatment in patients with moderate to severe plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable moderate to severe plaque-type psoriasis involving ≥5% body surface area
* History of plaque psoriasis for a minimum of 6 months prior to screening
* Age 18 - 75
* Males or females, females must be of non-childbearing potential (6 months post-menopausal, surgically sterilized) or using an approved form of birth control (oral contraceptives, Norplant®, Depo-Provera®, intrauterine device (IUD), double-barrier) and have a negative serum pregnancy test upon screening (Visit 1) and a negative urine test prior to randomization (Visit 2) into the trial
* Give informed consent and sign an approved consent form prior to any study procedures, including washout of prohibited medications

Exclusion Criteria:

* Primary guttate, erythrodermic, or pustular psoriasis
* Psoriasis which has failed to improve significantly with systemic treatments such as cyclosporine or methotrexate. Patients resistant to one, but have had a documented response to another may be included with approval of the medical monitor. Treatment failure will not include failure to improve if a full course of treatment was unable to be completed due to adverse events, intolerance of the treatment or administrative reasons
* Patients who have experienced treatment failure with a TNF-blocking agent. Treatment failure is defined as not achieving at least a 40% reduction in PASI score or having the TNF-blocking agent discontinued due to lack of efficacy
* Patients unable to wash out of all current psoriasis treatments (systemic, topical and phototherapy) except emollients and shampoos prior to beginning trial medication
* Patients taking the following medications known to elevate liver enzymes who have not been taking these medications at a stable dose for at least 1 month (3 months for diclofenac) without changes to liver functions tests (LFTs) prior to randomization (Visit 2): estrogens, oral contraceptives, selective serotonin reuptake inhibitors (SSRIs), nonsteroidal anti-inflammatory drugs (NSAIDs), acetominophen ≤3 g/day, aspirin, vitamin supplements (at recommended daily allowance doses). Patients taking doses of acetaminophen greater than three grams per day are excluded. Any other medication known to elevate hepatic enzymes not listed above is excluded
* Patients using any of the medications listed in the protocol, without the appropriate washout period
* Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis if the abnormality defines a disease listed as an exclusion criterion. All patients with a serum glutamate oxaloacetate transaminase, serum glutamate pyruvate transaminase , alkaline phosphatase greater than 1.5 x upper limit of normal (ULN) or total bilirubin greater than 1.0 x ULN will be excluded regardless of the clinical condition. Patients with serum creatinine, white blood cell (WBC) count, amylase, lipase, prothrombin time (PT), partial thromboplastin time (PTT), D-dimer, fibrin degradation product (FDP) greater than 1.5 x ULN, or blood smear poikilocytes or schistocytes greater than 1.0 x ULN will also be excluded. Patients with hemoglobinuria or proteinuria greater than 1+ will be excluded. Hemoglobinuria must be confirmed as hematuria with finding of red blood cell (RBC) on microscopic examination. Hematuria in a menstruating female will not require exclusion but must be repeated after menses has cleared prior to entry. Repeat laboratory testing is allowed once at screening prior to excluding the patient, to avoid excluding patients with transient or erroneous abnormal laboratory values
* Any clinically significant psychiatric illness which may interfere with the patient's participation in the trial or ability to interpret the trial results
* History of cardiovascular, renal, neurologic, liver, immunologic or endocrine dysfunction if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with any history of heart failure, patients with a recent history (i.e., 1 year or less) of myocardial infarction or patients with any arrhythmia requiring drug therapy
* Any ECG value outside of the reference range of clinical relevance including, but not limited to, QTcB >480 ms, PR interval >240 ms, QRS interval >110 ms
* History of malignancy in the past 5 years except treated cutaneous squamous cell or basal cell carcinoma
* Any active immunodeficiency or active infection, or any serious infection (requiring hospitalization or IV/intramuscular antibiotics) in the past 3 months prior to screening. Patients testing positive to human immunodeficiency virus (HIV), hepatitis B or hepatitis C will be excluded
* History of prior tuberculosis infection or active tuberculosis, patients must have a negative skin test or chest x-ray within the past 6 months prior to screening (Visit 1)
* History of drug or alcohol abuse within the past 2 years, active drug or alcohol abuse, or patients who consume more than three alcoholic drinks per day
* Patients who have taken an investigational drug within one month (30 days) or six half lives (whichever is greater) prior to screening (Visit 1). Patients who have been treated with any investigational antibody or other biological agent within the past 3 months are excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2001-06; Primary Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline for the total Psoriasis Area and Severity Index (PASI) score | after 4 weeks of treatment
Percent change from baseline for pathological thickness | after 4 weeks of treatment
Percentage of K16 negative assessments | at week 4
Number of patients with adverse events | up to 120 days
Number of patients with clinically significant effects on laboratory values | up to 36 days
Number of patients with abnormal findings in electrocardiogram | up to day 29
Number of patients with clinically significant changes in vital signs | up to day 36

SECONDARY OUTCOMES:
Absolute change from baseline in the number of epidermal T cells | after 4 weeks of treatment
Absolute change from baseline in the number of dermal T cells | after 4 weeks of treatment
Relative (%) change from baseline in the number of dermal T cells | after 4 weeks of treatment
Relative (%) change from baseline in the number of epidermal T cells | after 4 weeks of treatment
PASI 50 responder | after 4 weeks of treatment
  reduction of total PASI score by 50% or more
Assessment of target lesions on a 5-point numeric scale | day 1 and 29
Quantitative reverse transcriptase polymerase chain reaction (RT-PCR) gene expression for cytokines | days 1, 8 and 29
Reduction of serum immunological markers of disease activity | day 1 and 29
Change in score of total body lesion | day 1 and 29
Reduction of inducible nitric oxide synthase (iNOS) | day 1 and 29
PASI 75 responder | after 4 weeks of treatment
  reduction of total PASI by 75%
Histopathological global assessment on a 4-point scale | after 4 weeks of treatment
Keratin K16 improvement score | after 4 weeks of treatment
20% reduction responder variable for pathological thickness | after 4 weeks of treatment
20% reduction responder variable for iNOS | after 4 weeks of treatment
Reduction of K16 mRNA | day 1 and 29
Reduction of COX-2 mRNA | day 1 and 29
20% reduction responder variable for K16 | after 4 weeks of treatment
20% reduction responder variable for interleukin 8 mRNA | after 4 weeks of treatment